CLINICAL TRIAL: NCT02024815
Title: Comparable Investigation of One Fraction Radiotherapy (8 Gy x 1) and Multifraction Radiotherapy (3 Gy x 10) of Painful Bone Destructions in Patients With Multiple Myeloma.
Brief Title: Comparable Investigation of One Fraction Radiotherapy and Multifraction Radiotherapy in Patients With Multiple Myeloma.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Arturas Inciura, Prof., Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MM81310
Record Dates: First submitted 2013-12-19; First posted 2013-12-31 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Multiple Myeloma and Malignant Plasma Cell Neoplasms
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- External Beam radiotherapy (Experimental): Single 8 Gy fraction
  Interventions: Radiation: External Beam radiotherapy
- 3 Gy x 10 fractions (Active Comparator): External Beam radiotherapy - total dose 30 Gy, 3 Gy per fraction.
  Interventions: Radiation: External Beam radiotherapy

INTERVENTIONS:
Radiation: External Beam radiotherapy — External Beam radiotherapy

SUMMARY:
Radiotherapy is required to overcome pain and to evoke recalcification in multiple myeloma (MM) patients. Approximately 70% of all MM patients receive one or more radiotherapies in the course of their illness. The relief of pain is obtained in 75 - 100%. Recalcification is achieved in 40 - 50% of the irradiated bone destructions.There were a lot of randomized trials showed the same effect of single (SF) and multiple fractions (MF) in pain relief and recalcification for patients with painful bone metastases from solid tumors. The role of different palliative radiotherapeutic regimens for MM is not well established due to lack of clinical trials. Our prospective study analyzed the effect of two different radiotherapeutic regimens in the treatment of MM on pain relief, analgesics consumption and recalcification.

DETAILED DESCRIPTION:
The primary aim of our prospective study is to analyzed the effect of two different radiotherapeutic regimens in the treatment of MM on pain relief, the secondary aim is to analyzed the effect of two different radiotherapeutic regimens in the analgesics consumption and recalcification.

Eligibility criteria are age more than 18 years, Karnofsky index more than 40%, patients with painful bone destructions, patients with impending fracture in the region of destructions.

Exclusion Criteria are: patients with bone metastases from solid tumors, patients with solitary plasmacytoma, patients who had received previous irradiation to the present painful destruction site, patients who were incapable to complete the quality of life questionnaires, patients with poor health status.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky index more than 40%
* Patients with painful bone destructions.
* Patients with impending fracture in the region of destructions

Exclusion Criteria:

* Patients with bone metastases from solid tumors
* Patients with solitary plasmacytoma
* Patients who had received previous irradiation to the present painful destruction site,
* Patients who were incapable to complete the quality of life questionnaires
* Patients with poor health status .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-09; Primary Completion 2013-09 (Actual); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
To analyzed the pain relief in visual analogue scalewith the scale endpoints from 0 to 10 of two different radiotherapeutic regimens. | At admission and after 4, 12 and 24 weeks after radiotherapy

SECONDARY OUTCOMES:
To analyzed the analgesics consumption in two different radiotherapeutic regimens arms. | At admission and after 4, 12 and 24 weeks after radiotherapy

OTHER OUTCOMES:
To analyzed the recalcification on X rays in two different radiotherapeutic regimens arms. | At admission and after 4, 12 and 24 weeks after radiotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology Institute of Lithuanian of Health Sciences, Kaunas, Lithuania